CLINICAL TRIAL: NCT04218240
Title: Combining Pregabalin (LYRICA®) With Lofexidine (LUCEMYRATM): Can it Increase the Success of Transition to Naltrexone?
Brief Title: Combining Pregabalin (LYRICA®) With Lofexidine (LUCEMYRATM) to Treat OPIOID Withdrawal
Acronym: PGB-LOF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Kyle Kampman, Professor Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1UG3DA049694-01 (NIH)
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Opioid Withdrawal
MeSH Terms: interventions — Pregabalin; lofexidine

STUDY DESIGN:
Intervention Model Description: for the primary comparison of longitudinal subjective withdrawal measures, comparing the groups on rate of decrease across detox days, using a linear group by time effect for the mixed effects models described above. We have one primary outcome, so use an alpha level of 0.05, and we use two-sided tests. 90 subjects, 30 from each of three sites, who will be randomized into two groups, with 30 assigned to Lofexidine plus Placebo, and 60 to Lofexidine plus a starting daily dose of 400 mg of pregabalin and increasing to 600mg Pregabalin on day 2.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Penn Investigational Drug Service (IDS) will prepare blinded pregabalin capsules by over encapsulation of the drug into capsules shells matching the placebo capsules. Blinded pregabalin capsules will be packaged into blister packs along with lofexidine tablets, in separate compartments that are labeled for dosing times on days 1-7 and ship them to the research sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PGB/LFX; (Experimental): 0.54 mg lofexidine and 200 mg Pregabalin on days 1 -7 with taper for pregabalin and lofexidine starting on day 5
  Interventions: Drug: Pregabalin 200 MG capsules; Drug: Lofexidine 0.18Mg Tab
- Lofexidine and PLACEBO (Active Comparator): 0.54 mg lofexidine and Placebo (PLB) on days 1-7 with taper for lofexidine starting on day 5
  Interventions: Drug: Placebo oral tablet; Drug: Lofexidine 0.18Mg Tab

INTERVENTIONS:
Drug: Pregabalin 200 MG capsules — oral pregabalin 200 mg capsules given with a taper on day 5
  Other Names: lyrica
  Arms: PGB/LFX;
Drug: Placebo oral tablet — oral Placebo
  Arms: Lofexidine and PLACEBO
Drug: Lofexidine 0.18Mg Tab — lofexidine 0.18 tab given with a taper starting on day 5
  Other Names: lucemyra

SUMMARY:
A phase II double-blind placebo-controlled parallel group clinical trial that will randomize 90 subjects to investigate whether pregabalin (PGB) combined with Lofexidine (LFX) can reduce opioid withdrawal-related subjective effects, and investigate, whether the PGB/LFX combination can increase the proportion of patients with an opioid use disorder (OUD) who complete detoxification and transition to antagonist treatment with extended-release injectable naltrexone (XR-NTX).

DETAILED DESCRIPTION:
An inpatient detoxification study where pregabalin (PBG) will be given orally at a starting dose of up to 600 mg daily (group 1) tapered to 100 mg daily over 7 days; given with lofexidine (LFX) starting at 2.16 mg daily and declining to 0.72 mg over 7 days. On day 8, subjects are offered an injection of XR-NTX if they provide a urine sample that is negative for opioids and buprenorphine and pass a naloxone challenge. All subjects, regardless of whether or not they receive XR-NTX, will be given a referral and appointment for follow-up treatment when they leave the inpatient detoxification program.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects ≥ 18 years of age
2. Meet DSM-5 criteria for an Opioid Use Disorder with physiologic features. Have 2 or more of the 11 DSM 5 criteria for opioid disorder including tolerance and withdrawal features in the last 12 months
3. Interested in opioid antagonist treatment
4. Have used opioids in 20 or more of the last 30 days
5. Have a stable address in the local area; not planning to move; have documents for ID check
6. Absence of medical or psychiatric conditions that are likely to interfere with study participation
7. Have a 12 lead ECG demonstrating a QTc ≤450 msec and a QRS interval ≤120 msec. The site PI has the final determination for inclusion into the study for ECGs unless there is a question of QT prolongation or other factors (QTc/Fre uses the Frederica formula (QTc = QT/RR(1/3)). If consultation is needed, the PENN cardiologists and the medical monitor should be contacted
8. If female, have a negative pregnancy test and uses adequate contraception if of childbearing potential

Exclusion Criteria:

1. Current psychotic disorder (bipolar I, schizophrenia, major depression with psychotic features,) as defined by the MINI
2. An alcohol, benzodiazepine, or other sedative use disorder with physiological features that require medication for detoxification
3. History of allergy or other serious adverse event due to treatment with pregabalin, XR-NTX, or lofexidine
4. Pending incarceration in the next 30 days
5. Homicidal or otherwise behaviorally disturbed requiring immediate attention.
6. High Risk for suicide as determined by answering 'yes' to questions 4 and/or 5 on C-SSRS at screening
7. Blood pressure <90 mm Hg (systolic) or <60 mm Hg (diastolic). If this value is out of normal range, the investigator and a study clinician will decide subject inclusion or exclusion on a case-by-case basis
8. Heart rate and/or pulse<50 bpm at screening-sitting
9. An Estimated Glomerular Filtration Rate eGFR<90 mL/min/1.73m2
10. A History of, or current Seizure disorder (excluding childhood febrile seizures)
11. Inability to read and/or understand English. For example, unable to understand the informed consent as demonstrated by failing to answer 9/10 questions correctly on the quiz
12. Pregnant or breastfeeding
13. Currently taking sympathomimetic drugs, or a thiazolidinedione antidiabetic
14. An ALT and/or AST test that is at >4X the top limit of normal
15. A Child-Pugh score >7
16. Currently receiving opioids for pain management
17. In a treatment study where medication was administered in the last 30 days
18. Currently using medications that are known to be strong or moderate inhibitors of CYP2D6 such as fluoxetine, paroxetine, mirabegron, bupropion, quinidine, terbinafine, cimetidine, cinacalcet, duloxetine, or fluvoxamine
19. In a methadone maintenance or buprenorphine treatment program within the last 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Watson, Study Director — Office of Research Administration, Univ. of Pennsylvania
Locations (3):
- United States (3):
  - Mountain Manor Treatment Center, Baltimore, Maryland
  - John Mariani, New York, New York
  - Treatment Research Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Not at this time

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on media advertising from 3 treatment programs between December 2020 and March 2023. The first participant was enrolled on December 17, 2020 and the last participant was enrolled on 3/1/2023.
Pre-assignment Details: 90 consented and enrolled participants who met inclusion criteria and were randomized 1:1 ratio of either active pregabalin + lofexidine, or placebo pregabalin + lofexidine.
Groups:
- PGB/LFX;: oral tablet-lofexidine-active; oral capsule pregabalin-active Day 1: 0.54 mg lofexidine 3 times/day starting at 12p; plus 100 mg Pregabalin starting at 12p, and 4p, 200 mg at 8p. Day 2 through 5: 0.54 mg of lofexidine 4 times/day starting at 8a; plus 200 mg of pregabalin starting at 8am, 100 mg at 12p and 4p; and 200 mg at 8p.
  Taper starts on Day 5 for lofexidine at 0.54 at 8a, 0.36 at 12p, 4p and 8p plus pregabalin starting at 8am at 100 mg, 75 mg at 12p, 4p, and 150 at 8p.
  Taper on Day 6 for lofexidine at 0.36 at 8a, and 0.18 at 12p, 4p and 8p plus pregabalin starting at 8am at 50 mg, 25 mg at 12p, 4p, and 100 at 8p.
  Taper on Day 7 for lofexidine at 0.18 mg at 8a; 12p; 4p and 8p plus pregabalin at 25 mg; 8am,12p, 4p, and 8p.
- Lofexidine and PLACEBO: oral tablet-lofexidine-active; oral capsule pregabalin-placebo Day 1: 0.54 mg lofexidine 3 times/day starting at 12p; plus 100 mg Pregabalin-placebo starting at 12p, and 4p, 200 mg at 8p. Day 2 through 5: 0.54 mg of lofexidine 4 times/day starting at 8a; plus 200 mg of pregabalin-placebo starting at 8am, 100 mg at 12p and 4p; and 200 mg at 8p.
  Taper starts on Day 5 for lofexidine at 0.54 at 8a, 0.36 at 12p, 4p and 8p plus pregabalin-placebo starting at 8am at 100 mg, 75 mg at 12p, 4p, and 150 at 8p.
  Taper on Day 6 for lofexidine at 0.36 at 8a, and 0.18 at 12p, 4p and 8p plus pregabalin-placebo starting at 8am at 50 mg, 25 mg at 12p, 4p, and 100 at 8p.
  Taper on Day 7 for lofexidine at 0.18 mg at 8a; 12p; 4p and 8p plus pregabalin-placebo at 25 mg; 8am,12p, 4p, and 8p.
Period: Overall Study
Arm/Group | PGB/LFX; | Lofexidine and PLACEBO
Started | 58 | 32
Completed | 24 | 11
Not Completed | 34 | 21
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Lack of Efficacy | 24 | 19
Not completed — Physician Decision | 0 | 1
Not completed — Not Dosed Never met WD criteria | 4 | 1

BASELINE CHARACTERISTICS:
Population: males and females who are 18+ years of age, opioid use disorder
Groups:
- Total: Total of all reporting groups
Arm/Group | PGB/LFX; | Lofexidine and PLACEBO | Total
Number analyzed (Participants) | 58 | 32 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4138 (10.40417) | 37.6563 (10.2189) | 38.7889 (10.3157)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 45 | 24 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 54 | 32 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 32 | 23 | 55
  More than one race | 10 | 2 | 12
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 58 | 32 | 90
Fentanyl Use [Count of Participants; unit: Participants] — count of positive fentanyl urine results at baseline stratified by treatment
  Participants | 53 | 30 | 83

OUTCOME MEASURES:

1. Primary Outcome: Subjective Opioid Withdrawal Scale-Gossop (SOWS) Scale Score
Description: mild = 1-10 moderate=11-20 severe=21-30 higher number equals worse score
Time Frame: 7 days
Population: males, females 18+ years of age, opioid use disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PGB/LFX; | Lofexidine and PLACEBO
Number analyzed (Participants) | 58 | 32
score on a scale | 7.0 (4.6) | 9.1 (5.1)
Statistical Analysis 1: Comparison: PGB/LFX; vs Lofexidine and PLACEBO; A nonparametric (Kruskal-Wallis) comparison of the two groups (p=0.049); Test type: Superiority; p = .05, Chi-squared; 1 degree of freedom

2. Secondary Outcome: Completion of Withdrawal Management
Description: proportion of participants who completed the 7-day detoxification
Time Frame: 7 days
Population: male, females 18+ years of age, opioid Use diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | PGB/LFX; | Lofexidine and PLACEBO
Number analyzed (Participants) | 58 | 32
Participants
  completed detox | 23 | 9
  did not complete detox | 35 | 23
Statistical Analysis 1: Comparison: PGB/LFX; vs Lofexidine and PLACEBO; hypothesis: more people in active PGB/LFX will complete withdrawal CI = 95% P = 0.5; Test type: Other — Chi-square analysis; p = 0.27, Chi-squared

ADVERSE EVENTS:
Time Frame: 15 days per subject
Description: Withdrawal, unless clinically excessive is not considered an adverse event. Otherwise, definition is universal.
Arm/Group | PGB/LFX; | Lofexidine and PLACEBO
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/58 | 1/32
Other Adverse Events (participants affected / at risk) | 36/58 | 26/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PGB/LFX; (N=58) | Lofexidine and PLACEBO (N=32)
nausea with vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PGB/LFX; (N=58) | Lofexidine and PLACEBO (N=32)
bradycardia (Vascular disorders) | 10 (12) | 7 (9)
dizziness (Nervous system disorders) | 8 (8) | 8 (8)
orthostatic hypotension (Cardiac disorders) | 31 (64) | 20 (42)
sedation (Nervous system disorders) | 12 (13) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT04218240/Prot_SAP_002.pdf